CLINICAL TRIAL: NCT05742139
Title: Impact Sur la qualité de Vie et symptômes Persistants Des Patients à Distance d'Une neuroborréliose diagnostiquée et traitée
Brief Title: Impact on the Quality of Life and Persistent Symptoms of Patients Away From Diagnosed and Treated Neuroborreliosis
Acronym: QoLyme
Status: Completed | Type: Observational
Sponsor: Hopital Nord Franche-Comte (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-A01583-40
Record Dates: First submitted 2022-12-28; First posted 2023-02-23 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-10

CONDITIONS: Neuroborreliosis, Lyme; Quality of Life
MeSH Terms: conditions — Lyme Neuroborreliosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient group: Have been hospitalized or consulted for neuroborreliosis between 2010 and 2021; Have a diagnosis of probable neuroborreliosis (compatible clinical signs + lumbar puncture with positive intrathecal synthesis of immunoglobulins) or certain (compatible clinical signs + lumbar puncture with pleocytosis and positive intrathecal synthesis of immunoglobulins); Have received adequate treatment according to the recommendations (1st intention DOXYCYCLINE 100mgx2/day or 2nd intention CEFTRIAXONE IV 2g/day for 14 to 21
  Interventions: Other: Non intervention
- Control group: Be part of the entourage of the cases; Do not have ATCD of Lyme borreliosis (especially erythema migrans); Not having been bitten by a tick in the last 5 years;
  Interventions: Other: Non intervention

INTERVENTIONS:
Other: Non intervention — Non intervention

SUMMARY:
The link between Lyme neuroborreliosis (NBL) and persistent symptoms is debated in the medical world. Some report a frequency of post NBL symptoms similar to the general population, and others define a specific entity, the PTLDS (Post Treatment Lyme Disease Symptoms).

In France, few studies have evaluated the persistent symptoms and the impact on the quality of life of patients after treatment for NBL.

ELIGIBILITY:
Inclusion Criteria:

* Have been hospitalized or consulted for neuroborreliosis between 2010 and 2021;
* Have a diagnosis of probable neuroborreliosis (compatible clinical signs + lumbar puncture with positive intrathecal synthesis of immunoglobulins) or certain (compatible clinical signs + lumbar puncture with pleocytosis and positive intrathecal synthesis of immunoglobulins);
* Have received adequate treatment according to the recommendations (1st intention DOXYCYCLINE 100mgx2/day or 2nd intention CEFTRIAXONE IV 2g/day for 14 to 21

Exclusion Criteria:

* Be part of the entourage of the cases;
* Do not have ATCD of Lyme borreliosis (especially erythema migrans);
* Not having been bitten by a tick in the last 5 years;

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A online questionnaire is completed by the patient concerning socio-demographic date, patient history, quality of life scale, persistent neurological symptoms
Sampling Method: Non-Probability Sample
Enrollment: 159 (Actual)
Dates: Start 2023-02-27 (Actual); Primary Completion 2023-08-24 (Actual); Study Completion 2023-10-27 (Actual)

PRIMARY OUTCOMES:
Assess the quality of life of patients compared to a healthy control population using the SF-36 questionnaire and the Fatigue Scale Severity | At inclusion
Identification of symptoms recognized by the patient as persistent after neuroboreliosis from a list of referenced symptoms | At inclusion

SECONDARY OUTCOMES:
Imputability according to the patient of his pain in relation to the initial infection | At inclusion
Comparison of symptoms and/or quality of life between patients with definite versus probable neuroborreliosis using the SF-36 questionnaire | At inclusion

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU Besançon, Besançon
  - Hôpital Nord Franche-Comté, Trévenans

IPD SHARING:
Plan to Share IPD: No